CLINICAL TRIAL: NCT02412462
Title: A Phase I Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AB-16B5 in Subjects With an Advanced Solid Malignancy
Brief Title: Phase I Dose Escalation Study of AB-16B5 in Subjects With an Advanced Solid Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alethia Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-16B5-101
Record Dates: First submitted 2015-03-30; First posted 2015-04-09 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2016-07

CONDITIONS: Solid Tumor; Metastatic Cancer
Keywords: Phase I; Clusterin; Epithelial-to-Mesenchymal Transition (EMT); Circulating Tumor Cells (CTC); EMT and Stem Cell Biomarkers; Pharmacokinetics
MeSH Terms: conditions — Neoplasm Metastasis; Neoplastic Cells, Circulating

ARMS (1):
- AB-16B5 (Experimental): Single-arm study of AB-16B5 given as a 60-minute intravenous weekly infusion. One cycle of treatment will consist of 21 days. The dose levels that will be assessed are 1.5, 3.0, 6.0, 9.0 and 12 mg/kg.
  Interventions: Drug: AB-16B5

INTERVENTIONS:
Drug: AB-16B5

SUMMARY:
This is a Phase 1 clinical study to investigate the safety, pharmacokinetics and pharmacodynamics of AB-16B5 in patients with an advanced solid malignancy. AB-16B5 is a humanized monoclonal antibody that inhibits the activity of the secreted form of clusterin (sCLU), a potent inducer of the epithelial-to-mesenchymal transition (EMT). Eligible subjects will have a disease that has been refractory to prior therapy and is unlikely to benefit from known therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histologically or cytologically confirmed advanced solid malignancy that has been refractory to prior therapy and is unlikely to benefit from known therapies.
* Subjects may have measurable or non-measurable but evaluable disease.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 and an estimated life expectancy of at least 12 weeks.
* Subjects must be ≥ 18 years old.
* Male, or female subjects who are post-menopausal (amenorrheic for at least 12 months), or surgically or biologically sterile. Females of childbearing potential with a negative serum pregnancy test prior to entering the study and using adequate forms of contraception for the duration of the study, including 30 days after the last treatment. Males should avoid fathering children during the course of the study, and adequate methods of contraception should be used by both male and female subjects. Subjects and their partners with reproductive potential must use an effective contraceptive method while the subject is on the study treatment and for 30 days after the last treatment.
* Subjects must have adequate organ and immune function as indicated by the following laboratory values:

  * ANC ≥ 1.5 X 109/L
  * Platelets > 100 X 109/L
  * Hemoglobin ≥ 90 g/L
  * Serum creatinine ≤ 132 µmol/L
  * Total Bilirubin ≤ 1.5 X ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 X ULN* or;

    * 5 X ULN* (if hepatic metastases present)

      * ULN: Institution's upper limit of normal
* Subjects enrolled in the standard dose escalation portion of the study must have a tumor lesion amenable for biopsy with no contraindications for biopsy.
* Subjects must understand and be able and willing and likely to fully comply with the study procedures, including scheduled follow-up, and restrictions.
* Subjects must have given written personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines, before completing any study related procedures.

Exclusion Criteria:

* Subjects with medical, social, or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.
* Prior cancer therapy including surgery, radiotherapy, chemotherapy, hormonal and biological therapies within 3 weeks prior to study treatment.
* Uncontrolled brain metastases.
* Uncontrolled infection.
* Clinically significant ECG abnormalities.
* Known hypersensitivity of Grade > 2 to previous monoclonal antibody therapy.
* History of alcohol or other substance abuse within the last year.
* Use of another investigational agent in a clinical trial within the last 4 weeks prior to study treatment.
* Female subjects who are pregnant or lactating, including females with a positive pregnancy test at screening must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with an adverse event as a measure of safety and tolerability | Up to treatment discontinuation + 30 days with an estimated treatment duration of 6 to 24 weeks

SECONDARY OUTCOMES:
Determination of plasma concentrations of AB-16B5 | Several time-points during Cycle 1 and Cycle 2 for a total of 6 weeks
Objective tumor responses in subjects with measurable disease according to RECIST | Up to treatment discontinuation + 30 days with an estimated treatment duration of 6 to 24 weeks
Monitoring of epithelial-to-mesenchymal (EMT) and stem cells biomarkers in peripheral blood circulating tumor cells and paired tumor biopsies | Up to treatment discontinuation + 30 days with an estimated treatment duration of 6 to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada